CLINICAL TRIAL: NCT04966221
Title: Functional and Structural Lung Imaging in Chronic Obstructive Pulmonary Disease
Acronym: FASTCOPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Jonathan Brooke, Clinical Research Fellow, University of Nottingham
Other Study IDs: 21048
Record Dates: First submitted 2021-07-07; First posted 2021-07-19 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Alpha 1-Antitrypsin Deficiency
Keywords: MRI; COPD; A1ATD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adult healthy volunteers: Adult healthy volunteers, age matched to patient volunteers. Will undergo a combination of functional and structural lung MRI scans.
  Interventions: Diagnostic Test: Lung MRI scan
- Adults with Chronic Obstructive Pulmonary Disease: Will undergo a combination of functional and structural lung MRI scans. Some participants in this cohort will have lung volume reduction (LVR) as part of their normal clinical care. These participants will be given the option to attend two study visits - one before and one after LVR.
  Interventions: Diagnostic Test: Lung MRI scan
- Adults with alpha-1-antitrypsin deficiency: Will undergo a combination of functional and structural lung MRI scans.
  Interventions: Diagnostic Test: Lung MRI scan

INTERVENTIONS:
Diagnostic Test: Lung MRI scan — Participants will have a combination of structural and functional lung MRI scans. These scans will involve lying in a conventional MRI scanner while free breathing and may include additional breathing manoeuvres such as temporarily holding breath.

SUMMARY:
This study aims to use novel proton-based MRI techniques to assess lung function and structure in healthy volunteers and patients with chronic obstructive pulmonary disease (COPD) and alpha-1-anti-trypsin deficiency (A1ATD). These novel MRI measures will be compared to matched contemporary clinical diagnostic tools, namely pulmonary function tests (PFTs) and computed tomography (CT) scans. MRI has the advantages of avoiding ionising radiation exposure (unlike CT scans) and can also provide regional measures of lung function (unlike PFTs which provide global measures of function). In addition, these MRI techniques do not require the use of any inhaled or injected contrast agents.

Some patients enrolled in this study will be undergoing a lung volume reduction (LVR) procedure as part of their normal clinical care. LVR is an intervention for patients with severe lung disease and hyperinflation. It is a palliative therapy that helps to reduce lung hyperinflation through insertion of small valves in the airway or surgical removal of parts of the lung. This can lead to improvements in symptoms such as breathlessness and improve exercise tolerance due to better functioning of the lung. In this study, we will explore how lung MRI measures can be used to assess patients before and after an LVR intervention.

This study will take place at the University of Nottingham in collaboration with Nottingham University Hospitals NHS Trust. The study will last for 3 years and participants will be asked to attend a screening visit (lasting up to 1 hour) and either one or two study visits (each lasting up to 3 hours).

DETAILED DESCRIPTION:
This is a single centre pilot study. The research team aims to recruit adult healthy volunteers and adult patient volunteers with COPD and A1ATD. We have used similar proton-based MRI techniques in healthy volunteers and people with other lung diseases and the MRI scans have been well tolerated.

All participants will be adults (both male and female) who can give informed consent and are able to undertake the study procedures. Potential participants who cannot have an MRI scan for safety reasons (e.g. have a pacemaker) will not be recruited. During study visits, all research activities will be observed by a member of the research team.

During the screening visit (following consent), the following information and measures will be taken:

Relevant past medical history, COPD assessment tool (questionnaire), height, weight, blood pressure and pulse oximetry.

During study visits, a combination of structural and functional lung MRI scans will be performed with the participant lying in the scanner. Participants will be asked to breathe normally during scans and may also be asked to perform breathing manoeuvres such as holding their breath temporarily.

The participants will be assigned unique codes, and their data will be anonymised. Participants' medical reports will only be accessed for study purposes and will be treated as confidential.

The investigators will aim to use the data to plan future studies, and the data from this study may contribute to publications and presentations. Participants will not be identified in any publications arising from the research. The data obtained will be published without any identifying information.

ELIGIBILITY:
Workstream 1 Inclusion criteria (Adult Healthy Volunteers)

* Male or female aged 18 years and over
* Capacity to give informed consent
* Normal blood pressure (systolic BP > 90 mmHg and diastolic BP >50 mmHg)
* Resting heart rate > 50bpm
* For women, negative urinary β-hCG at the screening and subsequent visits (where clinical uncertainty of pregnancy)
* Subject able to hold breath for 10 seconds
* Subject able to understand the requirements of the study and to cooperate with the study procedures
* Subject has normal lung function by spirometry criteria
* Smoking history of > 10 pack years of tobacco smoking

Workstream 1 Exclusion criteria (Adult Healthy Volunteers)

* Unsuitable for MRI scanning (e.g. have metal implants or pacemaker or contraindicated following questionnaire)
* Subject deemed unlikely to comply with instructions during imaging
* Subject not deemed fit enough to tolerate procedure
* Subject deemed unsuitable by clinical investigator for other reasons
* Abnormal spirometry

Workstream 2 Inclusion criteria (Adults with chronic obstructive pulmonary disease)

* Male or female aged 18 years and over
* Capacity to give informed consent
* Normal blood pressure (systolic BP > 90 mmHg and diastolic BP >50 mmHg)
* Resting heart rate > 50bpm
* For women, negative urinary β-hCG at the screening and subsequent visits (where clinical uncertainty of pregnancy)
* Subject able to hold breath for 10 seconds
* Subject able to understand the requirements of the study and to cooperate with the study procedures
* Diagnosis of COPD made by respiratory physician and confirmed by spirometry criteria (FEV1/FVC ratio < 0.7) and > 10 pack years of tobacco smoking.

Workstream 2 Exclusion criteria (Adults with chronic obstructive pulmonary disease)

* Unsuitable for MRI scanning (e.g. have metal implants or pacemaker or contraindicated following questionnaire)
* Acute illness considered to be of sufficient severity to prevent safe MRI scanning. In this instance, the subject will be invited to be rescreened > 4 weeks later.
* Subject deemed unlikely to comply with instructions during imaging
* Subject not deemed fit enough to tolerate procedure
* Subject deemed unsuitable by clinical investigator for other reasons

Workstream 3 Inclusion criteria (Adults with COPD due to alpha-1-antitrypsin deficiency - A1ATD)

* Male or female aged 18 years and over
* Capacity to give informed consent
* Normal blood pressure (systolic BP > 90 mmHg and diastolic BP >50 mmHg)
* Resting heart rate > 50bpm
* For women, negative urinary β-hCG at the screening and subsequent visits (where clinical uncertainty of pregnancy)
* Subject able to hold breath for 10 seconds
* Subject able to understand the requirements of the study and to cooperate with the study procedures
* Diagnosis of A1ATD (PiZZ or PiZ-) and either evidence of emphysema on a previous clinical CT scan or evidence of airways obstruction

Workstream 3 Exclusion criteria (Adults with COPD due to alpha-1-antitrypsin deficiency - A1ATD)

* Unsuitable for MRI scanning (e.g. have metal implants or pacemaker or contraindicated following questionnaire)
* Acute illness considered to be of sufficient severity to prevent safe MRI scanning. In this case, the subject will be rescreened >4 weeks later
* Subject deemed unlikely to comply with instructions during imaging
* Subject not deemed fit enough to tolerate procedure
* Subject deemed unsuitable by clinical investigator for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include up to 25 participants in each of the three workstreams:
  Workstream 1 - Adult healthy volunteers Workstream 2 - Adults with chronic obstructive pulmonary disease Workstream 3 - Adults with COPD due to alpha-1-antitrypsin deficiency - A1ATD
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
To acquire structural and functional proton-based lung MRI scans from patients with COPD and COPD due to A1ATD and produce baseline data for these groups to inform future clinical studies | 3 years
  To compare functional MRI outcomes with matched clinical physiological data (e.g. pulmonary function tests) To compare structural lung images with matched conventional imaging techniques done for clinical reasons (e.g. computed tomography) of the diaphragm and lungs

SECONDARY OUTCOMES:
To assess the ability of participants of each group to adhere to the protocols, thus informing the study design of future trials | 3 years
To assess any change of MR outcomes across study visits for those participants undertaking more than one MR scanning visit. | 3 years
To assess any change of MR outcomes across study visits for participants who undergo LVR | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Philip Brooke, Principal Investigator — The University of Nottingham; Zachary Peggs, Principal Investigator — The University of Nottingham
Locations (1):
- Sir Peter Mansfield Imaging Centre, University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No